CLINICAL TRIAL: NCT02425215
Title: Does Hyperbaric Oxygen Therapy (HBOT) Reduce Pain, Improve Depression and Impact on Patients' Quality of Life for Those Suffering From Late Radiation Tissue Injury?
Brief Title: HBOT Late Radiation Tissue Injury
Status: Terminated | Type: Observational
Why Stopped: Lack of resources to complete the study
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-7413
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Late Radiation Injury; Chronic Pain
Keywords: Hyperbaric Oxygen Treatment; Late radiation injury; Adult; Malignancy; Quality of Life; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Radiotherapy is a common treatment for many malignancies. Radiation-related complications developing months or years after radiation treatment are known as late radiation tissue injury (LRTI) and are estimated to effect 5%-15% of all long-term survivors who have received radiation.

Hyperbaric oxygen therapy (HBOT) is a well established treatment of LRTI. Most of the studies evaluating effect of HBOT on LRTI are focused on survival, resolution of tissue damage and improvement in LENT-SOMA scale. Very few studies have addressed effect of HBOT on pain in LTRI. Krahn and colleagues were the first to report the analgesic effect of HBOT in 3 cases of refractory pain in oncological patients with radiation soft tissue injury. Other studies showed significant improvement in pain intensity in patients with breast cancer and pelvic malignancies treated with HBOT for LTRI. In patients that had developed radiation- induced brachial plexopathy, HBOT elicited an increase in warm pain thresholds and a reduction in lymphoedema. A prospective case study of 16 patients with gynecological cancer found no changes with respect to pain and depression outcomes. A trial in patients with radiation induced proctopathy showed that 75% of patients with rectal pain had some improvement, although none experienced a complete resolution of pain symptoms.

There are several mechanisms by which HBOT may elicit analgesic effects. There is a growing body of evidence that HBOT's analgesic effect related to nitric oxide metabolism and endogenous opioid secretion. Furthermore, the inhibition of tumor necrosis factor alph (TNF-α), the production of substance P, and the modulation of serotonergic pathways have all demonstrated a modification in the pain response following HBOT. In animal studies HBOT decreased allodynia and hyperalgesia in different models of neuropathic and inflammatory pain. The long lasting antinociceptive effect of HBOT was found to be dose-dependent in non-injured tissues.

In human studies, HBOT decreased pain and edema and improved function in patients suffering from the complex regional pain syndrome, and improved pain scores and range of motion in patients with idiopathic femoral head necrosis. Women suffering from interstitial cystitis demonstrated a reduction in pelvic pain following weeks and months of HBOT treatment. In patients suffering from idiopathic trigeminal neuralgia HBOT produced a rapid reduction in symptoms and these effects were lasting for 6 months following treatment. HBOT was also found to be an effective treatment for cluster headaches and migraines and alleviated muscle and bone pains in patients with myofascial syndrome, fibromyalgia, and biphosphonate-related osteonecrosis of the jaw.

Based on the evidence presented above and HBOT's known analgesic effect in many conditions, the investigators designed this study with the objective to evaluate if HBOT reduces pain, improves depression and impacts on patients quality of life in patients suffering from late radiation tissue injury.

Study Design: Prospective observational study (n=300). Patients that have had radiation therapy for malignancy, developed late radiation injury and suffer from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had radiation therapy, developed late radiation tissue injury and are eligible for hyperbaric oxygen therapy.
* Pain ≥ 5 in any anatomic site with duration > 3 months

Exclusion Criteria:

* Patient refusal
* Patient inability to answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing hyperbaric oxygen therapy for delayed radiation tissue injury in the Hyperbaric Unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (11 point numeric rating scale, Brief Pain Inventory short form ) | 6 months post-treatment
  Pain will be assessed with the 11 point numeric rating scale (NRS; 0 = "no pain" to 10 = "unbearable pain").Patients will be asked to document their pain during the previous 24 hours daily upon awakening and immediately after the intervention. Daily and weekly mean pain scores and the proportion of responders, defined as patients with a ≥30% reduction in mean pain score from baseline to endpoint will be recorded.
  The Brief Pain Inventory short form will also be administered.

SECONDARY OUTCOMES:
Pain Disability (pain disability index) | 6 months post-treatment
  Will be measured using the pain disability index (PDI). The tool is valid and reliable instrument widely used to assess chronic pain patients in research and clinical settings.
Quality of Life Measurement (EORTC QLQ C30) | 6 months post-treatment
  Will be assessed with the European Organization for Research and Treatment of Cancer Quality of life Questionnaire (EORTC QLQ C30). The EORTC QLQ-C30 is a self administered questionnaire developed to assess the quality of life of cancer patients. It has been translated and validated into 81 languages and is used in more than 3,000 studies worldwide. It is composed of both multi-item scales and single item measures.These include 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties).
The Patient Global Impression of Change | 6 months post-treatment
  The scale has been recommended by Initiatives on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) to evaluate the efficacy of treatment in chronic pain trials. It assesses global response to treatment and uses a 7-point Likert scale that varies from 1 (very much improved) to 7 (very much worse).
Depression and Anxiety (Hospital Anxiety (HADS-A) and Depression (HADS-D) scale) | 6 months post-treatment
  Depression and anxiety will be assessed with the Hospital Anxiety (HADS-A) and Depression (HADS-D) scale, consisting of 14 items (7 each for anxiety and depression).
Pain medications | 6 months post-treatment
  Change of pain medications.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada